CLINICAL TRIAL: NCT03638362
Title: Effect of Tart Cherry Juice on Inflammation and Dyslipidemia in Overweight and Obese Humans
Brief Title: Tart Cherry Juice and Chronic Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Keith Martin, Research Assistant Professor, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 10015542
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: CVD; Diabetes; Inflammation
Keywords: obese; overweight; tart cherry juice
MeSH Terms: conditions — Diabetes Mellitus; Inflammation; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Crossover Assignment In this study, the investigators recruited at-risk individuals who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with MetS. In this 10-week placebo-controlled 2 x 2 crossover dietary intervention, the investigators randomized participants to consume 240 mL (8 ounces) daily of either placebo (artificial cherry-flavored, anthocyanin-free beverage) or authentic TCJ for 4 weeks, followed by a 2-week washout period, then consumption of the alternate beverage for 4 weeks. Subsequently, the investigators determined the effect of TCJ in at-risk participants on markers of inflammation, glycemia, and lipidemia.
Who Masked: Participant
Masking Description: Placebo beverage was selected from commercially available, artificially flavored and colored fruit punches (Great Value fruit punch, Bentonville, AR) to match a closely as possible the color (red) of the TCJ.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants randomized to consume either placebo beverage or tart cherry juice at beginning of the study followed by a 2 week washout then switch over to the alternate beverage. Approximately half of participants began study consuming placebo beverage and the other half TCJ.
  Interventions: Dietary Supplement: Placebo
- Tart cherry juice (TCJ) (Experimental): Participants randomized to consume either placebo beverage or tart cherry juice at beginning of the study followed by a 2 week washout then switch over to the alternate beverage. Approximately half pf participants began study consuming placebo beverage and the other half TCJ.
  Interventions: Dietary Supplement: Tart cherry juice

INTERVENTIONS:
Dietary Supplement: Placebo — Participants consumed placebo beverage for 4 weeks.
  Arms: Placebo
Dietary Supplement: Tart cherry juice — Participants consumed tart cherry juice (8 ounces; 240 mL) per day for four weeks.
  Arms: Tart cherry juice (TCJ)

SUMMARY:
In this study, the investigators recruited at-risk individuals (n=10) who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with Metabolic Syndrome (MetS). In this 10-week placebo-controlled 2 x 2 crossover dietary intervention, the investigators randomized participants (n=10) to consume 240 mL (8 ounces) daily of either placebo (artificial cherry-flavored, anthocyanin-free beverage) or authentic TCJ for 4 weeks, followed by a 2-week washout period, then consumption of the alternate beverage for 4 weeks. In this study, the investigators determined the effect of TCJ in at-risk participants on markers of inflammation, glycemia, and lipidemia.

DETAILED DESCRIPTION:
In this study, the investigators recruited at-risk individuals (n=10) who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with MetS. Participants were >18 years of age, not pregnant, not diabetic, with no unresolved infections or diseases (diabetes, CVD, IBD, cancer and liver disease), and nonsmokers. Histories of medication and dietary supplement use were collected and those taking anti-inflammatory or lipid-lowering medications were excluded. After enrollment, subjects were randomly assigned to consume daily either 240 mL (8 ounces) of authentic TCJ (R.W. Knudsen, Chico, CA) or a placebo beverage (commercial fruit punch; Great Value, Bentonville, AR) for 4 weeks. After a 2-week washout period, participants consumed the alternate beverage for 4 weeks in this 10-week 2x2 crossover, placebo-controlled dietary intervention. Subsequently, the investigators determined the effect of TCJ in at-risk participants on markers of lipidemia (HDL, LDL, triglycerides, VLDL, total cholesterol), glycemia (fasting insulin and glucose, HOMA, QUICKI, McAuley indirect indices), and inflammation (hsCRP, TNF-alpha, and ESR).

ELIGIBILITY:
Inclusion Criteria:

* This study was a 12-week 2 x 2 crossover, randomized, placebo-controlled dietary intervention in overweight and obese participants (BMI>25.0 kg/m2) who are more likely to exhibit >1 of the 5 risk conditions associated with metabolic syndrome (MetS). BMI was the minimal criterion for recruitment.

Exclusion Criteria:

* Participants were >18 years of age, not pregnant, not diabetic, with no unresolved infections or diseases (diabetes, CVD, IBD, cancer and liver disease), and nonsmokers. Histories of medication and dietary supplement use were collected and those taking anti-inflammatory or lipid-lowering medications were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08-21 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
TCJ and hsCRP | 4 weeks
  high-sensitivity C-reactive protein (hsCRP), a marker of inflammation

SECONDARY OUTCOMES:
fasting triglycerides | 4 weeks
  Blood lipid and risk factor for CVD

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Martin, PhD, MTox, Principal Investigator — Principal Investigator, School of Health Studies

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be available to relevant parties, e.g., investigators, recognized scientific bodies, etc. upon reasonable request within an adequate time frame. Emails may be directed to the Principal Investigator.
Supporting Information: Study Protocol